CLINICAL TRIAL: NCT01866306
Title: A Dose-Finding and Longitudinal Biomarker Study of Rhinovirus Challenge in Healthy Volunteers and Mild-Moderate Asthmatics to Evaluate the Safety and Use of a Human Rhinovirus Preparation in Developing High Dimensionality Phenotypes ("Handprints") for Asthma
Brief Title: A Study to Evaluate the Safety and Use of Human Rhinovirus in Healthy and Asthmatic Participants (MK-0000-218)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: U-BIOPRED Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-218; 2013-000618-39 (EudraCT Number)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Healthy 10 TCID50 (Part 1) (Experimental): Healthy participants were treated with 10 Tissue Culture Infective Dose 50 (TCID50) administered by spraying an atomized viral suspension of RV16UB into a single nostril.
  Interventions: Biological: RV16UB
- Healthy 100 TCID50 (Part 1) (Experimental): Healthy participants were treated with 100 TCID50 administered by spraying an atomized viral suspension of RV16UB into a single nostril.
  Interventions: Biological: RV16UB
- Healthy 1000 TCID50 (Part 1) (Experimental): Healthy participants were treated with 1000 TCID50 administered by spraying an atomized viral suspension of RV16UB into a single nostril.
  Interventions: Biological: RV16UB
- Asthmatic non-LABA 10 TCID50 (Part 1) (Experimental): Participants with mild to moderate asthma, not concomitantly treated with LABA, were treated with 10 TCID50 administered by spraying an atomized viral suspension of RV16UB into a single nostril.
  Interventions: Biological: RV16UB
- Asthmatic non-LABA 100 TCID50 (Part 1) (Experimental): Participants with mild to moderate asthma, not concomitantly treated with LABA, were treated with 100 TCID50 administered by spraying an atomized viral suspension of RV16UB into a single nostril.
  Interventions: Biological: RV16UB
- Asthmatic LABA 100 TCID50 (Part 1) (Experimental): Participants with mild to moderate asthma, concomitantly treated with LABA, were treated with 100 TCID50 administered by spraying an atomized viral suspension of RV16UB into a single nostril.
  Interventions: Biological: RV16UB; Drug: LABA
- Asthmatic non-LABA 100 TCID50 (Part 2) (Experimental): Participants with mild to moderate asthma, not concomitantly treated with LABA, were treated with 100 TCID50 administered by spraying an atomized viral suspension of RV16UB into a single nostril.
  Interventions: Biological: RV16UB

INTERVENTIONS:
Biological: RV16UB — RV16UB is administered by spraying an atomized viral suspension into a single nostril. Planned doses of RV16UB in Part 1 are 10 Tissue Culture Infective Dose 50 (TCID50), 100 TCID50, 1000 TCID50 and 10,000 TCID50.
Drug: LABA — Asthmatic participants were treated with LABA as part of their standard of care
  Arms: Asthmatic LABA 100 TCID50 (Part 1)

SUMMARY:
The purpose of this study is to establish the safety and tolerability of Unbiased Biomarkers for the Prediction of Respiratory Disease Outcomes (U-BIOPRED) human rhinovirus 16 (RV16UB) in healthy and asthmatic participants, and to identify an appropriate dosage of RV16UB in order to study biomarkers in asthmatic participants. The study is divided into 2 parts. Part 1 is a dose-finding study where healthy participants, and asthmatic participants, who were either treated or not treated with a class of long-acting beta antagonists (LABA) will be recruited to undergo nasal challenge with increasing doses of RV16UB. Part 2 is a biomarker study where mild to moderate asthmatics undergo challenge with the most appropriate dose of RV16UB identified in Part 1, based on tolerability and viral effects. .

ELIGIBILITY:
Inclusion Criteria:

Parts 1 and 2:

* have a Body Mass Index (BMI) between =< 35 kg/m^2 and > 17 kg/m^2
* female of childbearing potential is not pregnant and agrees to use 2 acceptable methods of birth control until 10 days after the last visit,; or female is of non-childbearing potential
* is a non-smoker, or has not smoked within prior 12 months, with a history of =< 10 pack-years

Part 1:

Either of the following:

* healthy (may have out-of season seasonal allergies)
* mild to moderate-asthmatic with a history of spontaneous or exertional wheezing; and with all of the following for > 4 weeks prior: daytime symptoms twice weekly or less, no activity limitation, no nocturnal symptoms, uses reliever treatment twice daily or less, with an unchanged asthma medication dose, and uses inhaled corticosteroid (ICS) at a stable dose-equivalent of =< 500 mcg/day fluticasone propionate

Part 2:

* mild to moderate-asthmatics only with a history of spontaneous or exertional wheezing; and with all of the following for > 4 weeks prior: daytime symptoms twice weekly or less, no activity limitation, no nocturnal symptoms, uses reliever treatment twice daily or less, with an unchanged asthma medication dose, and uses ICS at a stable dose-equivalent of =< 500 mcg/day fluticasone propionate
* had a mild change in symptoms associated with viral syndrome, leading to temporarily increased short acting beta agonist use or increased ICS dose within the past 5 years

Exclusion Criteria:

* has a history of severe or difficult to manage allergies (e.g. food, drug, latex)
* has a history of asthma-related ventilatory failure in adolescence or adulthood
* is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* has significant nasal septum deviation, nasal polyps or other nasal anatomical abnormality
* shares the same household or has intimate contact with an infant, pregnant or lactating woman, or immunosuppressed individual
* has a history or current evidence of any upper or lower respiratory tract infection within 6 weeks prior to baseline assessment
* had major surgery or lost 1 unit (500 mL) of blood within prior 4 weeks
* has participated in another investigational trial within the prior 10 weeks
* is pregnant or a nursing mother
* uses excluded prescription or non-prescription medications within 2 weeks prior to initial viral challenge and throughout the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2015-12-25 (Actual); Study Completion 2016-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female healthy participants, and participants with mild-moderate asthma between the ages of 18 and 55 years (inclusive) were enrolled in this trial.
Period: Overall Study
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 23
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 23
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 23 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (9.6) | 39.7 (11.4) | 31.7 (10.1) | 31.7 (8.9) | 32.0 (10.2) | 31.7 (9.5) | 28.9 (9.3) | 31.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 1 | 5 | 5 | 13 | 35
  Male | 4 | 2 | 1 | 5 | 1 | 1 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Healthy and Asthmatic Participants With Events of Clinical Interest (ECI) (Part 1)
Description: ECI are selected non-serious and serious adverse events which include the following: an overdose of Sponsor's product; requirement for systemic steroids to treat asthma exacerbation related to virus challenge; acute reaction to virus challenge, confirmed through repeat measurement and when considered potentially associated with administration of virus; specified vital sign findings within 4hr of challenge; specified symptom findings within 24hr of challenge; >20% decrease in Forced Expiratory Volume in 1 second (FEV1) relative to baseline within 4hr of challenge; dyspnea associated with drop in FEV1 (within 4hr of challenge) that is unresponsive to a bronchodilator rescue agent within 20 minutes; Grade 2+ deviation from normal values of liver-related laboratory parameters at any time between challenge and day 14.
Time Frame: Up to Day 24
Population: Participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of viral challenge, according to the underlying scientific model. Participants from Part 2 were not analyzed.
Measure: Number; unit: Participants
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 0
Participants | 1 | 0 | 0 | 0 | 0 | 0 |

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAE) (Parts 1 and 2)
Description: A SAE is any adverse event occurring at any dose or during any use of the Sponsor's product that: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing in-patient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event.
Time Frame: Up to Day 24
Population: Participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of viral challenge, according to the underlying scientific model.
Measure: Number; unit: Participants
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Asthmatic Participants Treated With a Viral Dose of 100 TCID50 With Challenge Induced Upper Airway Symptoms (Part 1)
Description: Asthmatic participants from Part 1 were treated with RV16UB virus at a dose of 100 TCID50, and challenge induced upper airway symptoms were monitored with a diary recording Jackson Cold Symptom Score (CSS). The CSS measures 8 cold symptoms, with each symptom scored from 0 (absent) to 3 (severe). The total score ranges from 0-24, with higher scores reflecting greater severity. The number of participants with a CSS score equal or greater than 3 for two days in a row are presented.
Time Frame: Day 1 up to Day 7
Population: Participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of viral challenge, according to the underlying scientific model. Healthy participants, asthmatics treated with a viral dose of 10 TCID 50, and participants from Part 2 were not analyzed.
Measure: Number; unit: Participants
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 6 | 0
Participants |  |  |  |  | 6 | 5 |

4. Primary Outcome: Time -Weighted Average (TWA) Percent Change From Baseline (CFB) in Morning FEV1 in Asthmatic Participants on Days 1-7 (Part 2)
Description: Log-transformed FEV1 data were fit by Bayesian hierarchical longitudinal models, with a random participant effect and a fixed categorical effect for day. All baseline (day -7 to day -1) FEV1 were assumed to be with equal mean. FEV1 assessments obtained between 3 am to 3 pm were counted as morning measurements. The TWA CFB morning FEV1 on days 1-7 was calculated as the difference of the mean of estimated day 1-7 morning FEV1 value and the corresponding estimated baseline value. The 95% Confidence Interval actually refers to a 95% Credible Interval. The anticipated mean reduction from baseline is 10%.
Time Frame: Baseline and Days 1 - 7
Population: Participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of viral challenge, according to the underlying scientific model. Participants from Part 1 were not analyzed; one participant who received a viral dose of 67 TCID50, was included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23
Percent change |  |  |  |  |  |  | -1.840 [-2.959 to -0.706]

5. Primary Outcome: TWA Percent CFB in Evening FEV1 in Asthmatic Participants on Days 1-7 (Part 2)
Description: Log-transformed FEV1 data were fit by Bayesian hierarchical longitudinal models, with a random participant effect and a fixed categorical effect for day. All baseline (day -7 to day -1) FEV1 were assumed to be with equal mean. FEV1 assessments obtained between 3 pm to next day 3 am were counted as evening measurements. The TWA CFB evening FEV1 on days 1-7 was calculated as the difference of the mean of estimated day 1-7 evening FEV1 value and the corresponding estimated baseline value. The FEV1 readings on the evenings of sputum inductions were excluded from the analyses. The 95% Confidence Interval actually refers to a 95% Credible Interval. The anticipated mean reduction from baseline is 10%.
Time Frame: Baseline and Days 1- 7
Population: Participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of viral challenge, according to the underlying scientific model. Participants from Part 1 were not analyzed; one participant who received a viral dose of 67 TCID 50, was included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23
Percent change |  |  |  |  |  |  | -2.134 [-3.321 to -0.943]

6. Primary Outcome: Change From Baseline in Mean Maximum Jackson Cold Symptom Score (CSS) on Days 1 to 14 in Asthmatic Participants (Part 1)
Description: Asthmatic participants from Part 1 were treated with RV16UB virus, and challenge induced upper airway symptoms were monitored with a diary recording CSS. The CSS measures 8 cold symptoms, with each symptom scored from 0 (absent) to 3 (severe). The total score ranges from 0-24, with higher scores reflecting greater severity, and a positive change from baseline indicating worsening symptoms.
Time Frame: Baseline and Days 1 - 14
Population: Participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of viral challenge, according to the underlying scientific model. Healthy participants, and participants from Part 2 were not analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 0
Score on a scale |  |  |  | 6.05 (3.18) | 6.99 (3.22) | 9.56 (4.76) |

7. Primary Outcome: Number of Asthmatic Participants Demonstrating at Least 10^3 Copies/ml of Viral RNA in Nasal Lavage Fluid on Days 1 to 14 (Part 1)
Description: Viral RNA was measured by real time reverse transcriptase polymerase chain reaction (qRT-PCR) from nasal lavage fluid collected on day 3 and day 7 from asthmatic participants, and the number of participants with at least 10^3 copies/ml was determined.
Time Frame: Days 1 - 14
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 0
Participants |  |  |  | 4 | 5 | 6 |

8. Secondary Outcome: Mean Percent Change From Baseline in Maximum Drop FEV1 of Asthmatic Participants (Part 2)
Description: Log-transformed FEV1 data were fit by Bayesian hierarchical longitudinal models, with a random participant effect and a fixed categorical effect for day. All baseline (day -7 to day -1) FEV1 were assumed to be with equal mean. The FEV1 readings on the evenings of sputum inductions were excluded from the analyses. The percent decrease of the lowest FEV1 measurement after viral challenge compared to the TWA of the baseline FEV1 is presented. The 95% Confidence Interval actually refers to a 95% Credible Interval. The mean percent decrease is anticipated to be different from zero.
Time Frame: Baseline and up to day 7
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23
Percent change |  |  |  |  |  |  | -6.838 [-9.316 to -4.835]

9. Secondary Outcome: Mean Change From Baseline in TWA Asthma Control Diary (ACD) Score of Asthmatic Participants on Days 3 to 10 (Part 2)
Description: The ACD contains seven symptom questions (nocturnal awakening, waking in the morning with symptoms, activity limitation, shortness of breath and wheezing) which are answered on rising in the morning and retiring at bedtime. Missing scores are imputed by linear interpolation or extrapolation. Daily ACD score was fit by a Bayesian hierarchical longitudinal model with participant-specific intercept and a fixed categorical effect for day. All baseline (day -7 to day -1) ACD scores are assumed to be with equal mean. The ACD score is the sum of responses to the seven questions, with answers on a 7-point scale (0= no impairment; 6 = maximum impairment) with the score ranging from 0 to 42, and higher scores indicating greater impairment. The 95% Confidence Interval actually refers to a 95% Credible Interval. The mean percent increase is anticipated to be different from zero.
Time Frame: Baseline and Days 3 to 10
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23
Score on a scale |  |  |  |  |  |  | 2.732 [2.282 to 3.177]

ADVERSE EVENTS:
Time Frame: Up to day 24
Description: Participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of viral challenge, according to the underlying scientific model.
Arm/Group | Healthy 10 TCID50 (Part 1) | Healthy 100 TCID50 (Part 1) | Healthy 1000 TCID50 (Part 1) | Asthmatic Non-LABA 10 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 1) | Asthmatic LABA 100 TCID50 (Part 1) | Asthmatic Non-LABA 100 TCID50 (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 1/6 | 0/23
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 4/6 | 0/6 | 2/6 | 5/6 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy 10 TCID50 (Part 1) (N=6) | Healthy 100 TCID50 (Part 1) (N=6) | Healthy 1000 TCID50 (Part 1) (N=6) | Asthmatic Non-LABA 10 TCID50 (Part 1) (N=6) | Asthmatic Non-LABA 100 TCID50 (Part 1) (N=6) | Asthmatic LABA 100 TCID50 (Part 1) (N=6) | Asthmatic Non-LABA 100 TCID50 (Part 2) (N=23)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy 10 TCID50 (Part 1) (N=6) | Healthy 100 TCID50 (Part 1) (N=6) | Healthy 1000 TCID50 (Part 1) (N=6) | Asthmatic Non-LABA 10 TCID50 (Part 1) (N=6) | Asthmatic Non-LABA 100 TCID50 (Part 1) (N=6) | Asthmatic LABA 100 TCID50 (Part 1) (N=6) | Asthmatic Non-LABA 100 TCID50 (Part 2) (N=23)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.